CLINICAL TRIAL: NCT03003780
Title: Mindful Steps: Coupling Technology and Mind-Body Exercise to Facilitate Physical Activity in Patients With Cardiopulmonary Disease
Brief Title: Mindful Steps: Promoting Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P000368
Record Dates: First submitted 2016-12-13; First posted 2016-12-28 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Copd; Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Steps (Experimental): Web-based behavioral intervention
  Interventions: Behavioral: Mindful Steps
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Mindful Steps — Integrated website, activity tracker, and mind-body training
  Arms: Mindful Steps

SUMMARY:
This is a developmental project with two phases. The first phase will adapt an existing web-based intervention to incorporate mind-body exercises to develop a multi-modal intervention to promote physical activity in patients with COPD and HF. The second phase will pilot test this new intervention in a longitudinal study (subjects randomized to intervention or usual care).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD OR clinical diagnosis of HF syndrome (New York Heart Association Class 1-3)
* Able to participate in an exercise program
* Have an active email account and access to a computer with internet connection

Exclusion Criteria:

* COPD or HF exacerbation in the previous month
* Inability to ambulate
* Clinical signs of unstable cardiovascular disease
* Hypoxemia during 6MWT
* Inability to collect at least 7 of 14 days of baseline step counts
* Current participation in a cardiac or pulmonary rehabilitation program.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  intervention acceptability (qualitative interview)

SECONDARY OUTCOMES:
Self-efficacy | baseline, months 3, 6, 9 and 12
  change in self-efficacy between time points (exercise self-efficacy scale)
Physical activity | baseline, months 3,6,9, and 12
  change in physical activity between time points (physical activity questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- BIDMC, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kraemer KM, Litrownik D, Wayne PM, Richardson CR, Bhomia N, Kadri R, Rist PM, Ngo L, Moy ML, Yeh GY. Promoting Walking in Cardiopulmonary Disease With Mindful Steps: Pilot Feasibility Randomized Controlled Trial of a Web-Based, Pedometer-Mediated Mind-Body Intervention. JMIR Form Res. 2025 Oct 28;9:e74118. doi: 10.2196/74118. PMID 41147625
- [Derived] Litrownik D, Gilliam EA, Wayne PM, Richardson CR, Kadri R, Rist PM, Moy ML, Yeh GY. Development of a Novel Intervention (Mindful Steps) to Promote Long-Term Walking Behavior in Chronic Cardiopulmonary Disease: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Apr 29;10(4):e27826. doi: 10.2196/27826. PMID 33913819